CLINICAL TRIAL: NCT07140172
Title: Axillary Radiotherapy or Axillary Lymph Node Dissection in Patients With Clinically Node- Positive Breast Cancer Undergoing Upfront Tailored Axillary Surgery: An International, Randomized Superiority Trial (OPBC-10/ NOAX)
Brief Title: Axillary Radiotherapy or Axillary Lymph Node Dissection in Patients With Clinically Node- Positive Breast Cancer Undergoing Upfront Tailored Axillary Surgery
Acronym: OPBC-10/ NOAX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01460; NOAX; bb24Weber2
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: axillary lymph node dissection (ALND); axillary radiotherapy (ART); tailored axillary surgery (TAS); clinically node positive breast cancer (cN+ BC); sentinel lymph node biopsy (SLNB); Breast cancer-specific survival (BCSS); NOAX; OPBC-10; Lymphedema; Quality of life (QoL)
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: International, multicenter, randomized controlled, superiority trial comparing TAS and ART (experimental group) to ALND (control group) in terms of arm-related QoL and occurrence of lymphedema two years after randomization (co-primary endpoints).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Control): ALND (Active Comparator): 1. Surgery: Tailored Axillary Surgery (TAS) includes the sentinel lymph node (SLN) procedure, radiographic confirmation of the removal of previously marked lymph nodes (clip removal), and the targeted excision of palpably suspicious lymph nodes.
  2. Surgery: ALND - current standard of care, with the intention to remove the entire soft tissue within the anatomical borders of the axilla.
  3. Radiotherapy: All patients receive adjuvant breast irradiation following breast-conserving surgery, along with extended regional lymph node irradiation (breast/chest wall irradiation excluding the axilla).
  Interventions: Procedure: Axillary lymph node dissection (ALND)
- Arm B (Investigational): ART (Active Comparator): 1. Surgery: Tailored Axillary Surgery (TAS) includes the sentinel lymph node (SLN) procedure, radiographic confirmation of the removal of previously marked lymph nodes (clip removal), and the targeted excision of palpably suspicious lymph nodes.
  2. Radiotherapy: All patients receive adjuvant breast irradiation following breast-conserving surgery, along with extended regional lymph node irradiation (breast/chest wall irradiation excluding the axilla).TAS + breast/chest wall and axillary irradiation (ART)
  3. Radiotherapy: Axillary radiotherapy (ART).
  Interventions: Procedure: Axillary radiotherapy (ART)

INTERVENTIONS:
Procedure: Axillary lymph node dissection (ALND) — Surgical removal of lymphatic tissue within the anatomical boundaries of the axilla (standard of care in the upfront surgery setting in patients with cN+ BC)
  Arms: Arm A (Control): ALND
Procedure: Axillary radiotherapy (ART) — Axillary irradiation
  Arms: Arm B (Investigational): ART

SUMMARY:
This trial is to investigate if in patients with clinically node positive breast cancer undergoing upfront surgery, treatment with TAS and ART is superior to ALND in terms of arm-related Quality of Life (QoL) and occurrence of lymphedema two years after randomization.

DETAILED DESCRIPTION:
Despite major morbidity, axillary lymph node dissection (ALND) is standard of care in patients with clinically node positive breast cancer (cN+ BC) who undergo upfront surgery, which is frequently indicated in case of luminal biology. Tailored axillary surgery (TAS) was shown to selectively target positive nodes, thereby removing significantly more nodes than sentinel lymph node biopsy (SLNB), but less nodes than ALND. Therefore, it is currently unclear if TAS in combination with axillary radiotherapy (ART) exposes the axilla to less harm compared to ALND. It is hypothesized that patient's quality of life (QoL) and morbidity can be improved by replacing ALND with the combination of TAS and ART in patients undergoing upfront surgery.

The main goal of this trial is to investigate if in patients with clinically node positive breast cancer undergoing upfront surgery, treatment with TAS and ART is superior to ALND in terms of arm-related QoL and occurrence of lymphedema two years after randomization.

ELIGIBILITY:
Inclusion Criteria at screening:

* Written informed consent according to ICH/GCP regulations prior to any trial specific procedures.
* Patients ≥ 18 years of age.
* Node-positive breast cancer (histologically or cytologically proven both in primary tumor and in lymph node) American Joint Committee on Cancer/ International Union Against Cancer (AJCC/UICC) stage II-III (all molecular subtypes allowed).
* Node-positivity detected by imaging and non-palpable (iN+) and confirmed by pathology.
* Node-positivity palpable (cN1-3) and confirmed by pathology.
* Occult breast cancer is allowed, if biopsy-proven axillary lymphatic metastasis is present.
* Eligible for primary ALND or SLN procedure and either:

  * Newly diagnosed.
  * Isolated in-breast recurrence or second ipsilateral breast cancer after previous breast conserving surgery and sentinel procedure and at least 3 years disease free and no prior axillary dissection or axillary RT.
* Upfront surgery setting.
* Most suspicious axillary lymph node clipped. (If clipping is not part of the routine, this should be done after consent of the patient as a study procedure.)
* Ability to complete the QoL questionnaires.
* WHO performance status 0-2
* Adequate condition for general anesthesia, breast cancer surgery and radiotherapy.
* Adult patients (≥18 years of age).
* Women of child-bearing potential are using effective contraception (condom, diaphragm, intrauterine device), are not pregnant or lactating and agree not to become pregnant during trial treatment (until end of RT) and thereafter during the time recommended by the guidelines - also for adjuvant systemic therapies. A negative pregnancy test before registration is required for all women of child-bearing potential.
* Men agree not to father a child during trial treatment and for 6 months afterward.

Exclusion criteria at screening:

* Stage IV breast cancer.
* Clinical N3c breast cancer without axillary disease (clinical N3a and clinical N3b are allowed).
* Clinical N2b breast cancer (clinical N2a is allowed).
* Contralateral breast cancer within 3 years.
* Prior axillary surgery (except prior sentinel node procedure in case of in-breast recurrence).
* Prior regional radiotherapy.
* Neoadjuvant treatment with the exception of bridging therapy given for less than 3 months.
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from pre-registration with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Exclusion criteria at randomization (intraoperatively):

* Absence of clip in the specimen radiography.
* Palpable disease left behind in the axilla after TAS.
* No SLN identified in the axilla.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Change in arm-related Quality of Life (QoL) | From baseline to 2 years after randomization
  The arm subscale (ARM) of the FACT-B+4 is used to assess arm-related QoL.The FACT-B comprises five subscales: physical well-being (seven items), social well-being (seven items), emotional well-being (six items), functional well-being (seven items), and concerns specific to patients with breast cancer (13 items). The FACT-B+4 questionnaire consists of the FACT-B subscales and the additional ARM subscale including five questions related to arm morbidity with four additional validated arm morbidity items that are added to the one item on arm morbidity already included in the FACT-B questionnaire. Patients are asked to indicate on a five- point scale from 0 (not at all), 1 (a little bit), 2 (somewhat), 3 (quite a bit), to 4 (very much), to what degree each statement applied over the previous 7 days. The individual scoring of each question is inverted and added up to the total score ranging between 0 and 20 points, higher scores representing less arm problems.
Occurrence of lymphedema | From baseline to 2 years after randomization
  Bilateral measurements will be obtained 10 cm above and 5 cm below the olecranon process on both the ipsilateral and contralateral upper extremities. The change in ipsilateral upper- extremity circumference, corrected for any change in the contralateral upper extremity, will be calculated using the following formula: L = (Ia - Ib) - (Ca- Cb).
  It indicates ipsilateral upper-extremity circumference, C indicates contralateral upper- extremity circumference, a indicates assessments during trial treatment and follow-up, and b indicates baseline assessment. L will be calculated for both upper arm and forearm, and lymphedema is defined as present if L > 2 cm for either location. The proportion of patients with lymphedema will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Walter P. Weber, Prof. Dr. med., Principal Investigator — Breast Surgery Service, University Hospital Basel
Locations (36):
- Duke University/Duke Cancer Center, Durham, North Carolina, United States
- Sanatorio Parque Breast Cancer Center, Rosario, Argentina
- Austria (3):
  - KH Dornbirn, Dornbirn
  - LKH Feldkirch, Feldkirch
  - MUI - Univ. Klinik f. Frauenheilkunde Innsbruck, Innsbruck
- CIUSSS du Centre Ouest-de-l 'Ile-de-Montréal, Montreal, Canada
- Croatia (2):
  - Breast Centre of Clinical Hospital, Rijeka, Rijeka
  - HRUHC Sestre milosdrnice, Zagreb, Zagreb
- Germany (2):
  - Brustzentrum Heidelberg Klinik St. Elisabeth GmbH, Heidelberg
  - HELIOS Universitätsklinikum Wuppertal, Wuppertal
- Greece (3):
  - "Alexandra" Hospital, Athens, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Larissa, Larissa
- Policlinico Universitario "Agostino Gemelli, Rome, Italy
- South Korea (2):
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Switzerland (18):
  - Kantonsspital Baden, Baden
  - Breast Surgery Service, University Hospital Basel, Basel
  - Clinique des Grangettes, Chêne-Bougeries
  - Spital Thurgau, Frauenfeld
  - Hôpitaux Universitaires de Genève, Geneva
  - Clinique de Genolier, Genolier
  - Hirslandenklinik St. Anna, Lucerne
  - Kantonsspital Luzern, Lucerne
  - Centro di Senologia della Svizzera Italiana, Lugano
  - Hôpital Neuchâtelois, Neuchâtel
  - Kantonsspital St. Gallen, Sankt Gallen
  - Tumor-& Brustzentrum Ostschweiz St. Gallen, Sankt Gallen
  - Spital Limmattal, Schlieren
  - Hôpital du Valais, Hôpital de Sion, Sion
  - Kantonsspital Winterthur, Winterthur
  - Spital Zollikerberg, Zollikerberg
  - Brustzentrum Zürich (Seefeld), Zurich
  - Stadtspital Triemli, Zurich
- Turkey (Türkiye) (2):
  - İstanbul Bağcılar Training and Research Hospital, Istanbul
  - Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, Istanbul